CLINICAL TRIAL: NCT04534010
Title: A Single Arm, Single Center Pilot Study Evaluating the Safety and Healing Time of a Decellularized, Whole Donor Nipple-Areola Complex Reconstruction Graft
Brief Title: Decellularized, Whole Donor Nipple-Areola Complex Reconstruction Grafts
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision due to low accrual
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Arash Momeni, Assistant Professor of Surgery, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-55153; BRS0117 (Other: OnCore)
Record Dates: First submitted 2020-08-20; First posted 2020-09-01 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- NACgraft patients (Experimental): uni- or bilateral engraftment surgery will be performed
  Interventions: Device: NACgraft

INTERVENTIONS:
Device: NACgraft — Patients requiring reconstruction of their nipple and areola have a NACgraft surgically implanted on their breasts. A NACgraft is a novel decellularized cadaveric implant derived from human nipples.

SUMMARY:
The goal of this study is to evaluate safety and healing time after nipple-areolar complex (NAC) reconstruction with the BioAesthetics' decellularized human nipple-areolar complex (dcl-hNAC) graft in patients who have had autologous breast reconstruction for breast cancer. Secondary objectives will be to assess patient satisfaction, patient well-being, patient self-esteem, patient body image, patient psychological well-being, nipple dimensions and sensitivity following NAC reconstruction surgery with the BioAesthetics' dcl-hNAC graft.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18-65
* Patient desires NAC grafting ≥3 months after autologous breast reconstruction
* Patient agrees to sleep on back until grafts healed (6 weeks)
* Patient agrees to abstain from aspirin, alcohol, or excessive caffeine until grafts healed (6 weeks)
* Patient agrees to not undergo NAC tattooing until completing study (12 months)
* Patient is able to understand and willing to sign informed consent.

Exclusion Criteria:

* History of delayed wound healing
* history of Vitamin C deficiency
* history of diabetes (Type I or Type II)
* current BMI<18.5 or >40 kg/m,
* patient has any other uncontrolled comorbidity.
* Patient has a history of allergic reaction to any decellularized biologic matrix product.
* Patient is currently smoking or using tobacco or nicotine products (i.e. patch, gum, or nasal spray) or has used such products in the past 12 months.
* Patient is currently receiving radiation or chemotherapy or received radiation to the breast wall.
* Patient has a history of prior NAC reconstruction
* Patient has had NAC tattooing.
* Patient is pregnant, breastfeeding or planning to become pregnant during the study period.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey C Gurtner, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: grafts
Groups:
- NACgraft patients: Patients requiring reconstruction of their nipple and areola have a NACgraft surgically implanted on their breasts.
Period: Overall Study
Arm/Group | NACgraft patients
Started | 6; 11 grafts
Completed | 4; 8 grafts
Not Completed | 2; 3 grafts

BASELINE CHARACTERISTICS:
Arm/Group | NACgraft Patients
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Grafts With Complete Healing
Description: Complete is defined as when the graft is >99% epithelialized. Degree of healing will be based on visual assessment by the surgeon and central reviewer with the following metrics on a visual analog scale (VAS): epithelialization (0-100%); granulation (0-100%); overall healing (0-100%). Photographs will be taken using a standardized 3d imaging device, stored and transmitted securely to a central reviewer for independent review.
Time Frame: 3, 6 and 12 months
Population: Participant who complete the protocol
Measure: Count of Units; unit: grafts
Units Other Than Participants: grafts
Arm/Group | NACgraft patients
Number analyzed (Participants) | 4
Number analyzed (grafts) | 8
grafts
  3 months | 8
  6 months | 8
  12 months | 8

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | NACgraft patients
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NACgraft patients (N=6)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Not related (due to preexisting metastatic breast cancer)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NACgraft patients (N=6)
Graft sloughing (Surgical and medical procedures) | 2 — Anticipated adverse effect

LIMITATIONS AND CAVEATS:
Early termination led to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT04534010/Prot_SAP_000.pdf